CLINICAL TRIAL: NCT06550635
Title: Joint and Hematologic Disorders of Noonan Syndrome: French Descriptive Cross-sectional Study (NOORHA)
Brief Title: Joint and Hematologic Disorders of Noonan Syndrome: French Descriptive Cross-sectional Study
Acronym: NOORHA
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: NOORHA (29BRC19.0038)
Record Dates: First submitted 2019-06-05; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2020-06

CONDITIONS: Noonan Syndrome
MeSH Terms: conditions — Noonan Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Noonan's syndrome is a rare genetic disease, estimated to be between 1: 1000 to 1: 2500 and characterized by cardiothoracic malformations, sometimes mental retardation, but also by hematologic abnormalities and joint involvement. These are poorly described in the literature. The aim of this work is therefore to describe the frequency and type of these manifestations in the French pediatric population and to compare patients with and without these disorders.

DETAILED DESCRIPTION:
Noonan Syndrome is a genetic disease whose prevalence is not clearly defined and would be between 1/1000 and 1/2500.

Affected patients have various morphological abnormalities, cardiothoracic malformations, sometimes mental retardation, but also haematological abnormalities and joint damage.

Diagnostic criteria have been proposed among which, the most used are van der Burgt's criteria.

Genetics is heterogeneous. A genetic abnormality can be found in 75% of cases. Affected genes encode proteins involved in the RAS / MAPK pathway (Mitogen Activated Protein Kinase), resulting in deregulation of this pathway. The latter is involved in several development processes determining morphotype, organogenesis, synaptic plasticity and growth.

There are also thoracic and abdominal deformities (upper pectus carinatum and inferior excavatum, large nipple spacing), spinal deformities in 30% of cases with a recommended correction in 2/3 of the cases. It is described ulna valgus and genuvalgum.

Concerning haematological disorders:

Children with Noonan Syndrome are predisposed to a number of hematologic abnormalities. The most common haematological lesions are coagulopathies caused by a deficiency of coagulation factors or platelet dysfunction that seem to affect one third of patients.

Concerning rheumatological disorders:

Hemophilias, due to recurrent bleeding, may develop secondarily hemophilic arthropathies.

There are several pediatric cases of granulomatous gigantocellular tumors and pigmented villonodular synovitis that are synovial proliferations affecting the joints, tendon sheaths and bursae. Villonodular synovitis is also a granulomatous giant cell lesion. Unlike villonodular synovitis in the general population, reported cases are frequently polyarticular. The diffuse villonodular synovitis in the general population has an estimated frequency of 1.8 cases per million. It is most often developed in adulthood (20-50 years), but can also begin in childhood.

There has been no description of arthritis or isolated arthralgia.

Regarding abnormalities of bone metabolism, even if there is a tendency to short stature, and there are bone dysplasias, little information is available regarding the mineralization and bone metabolism in Noonan syndrome. An increase in bone resorption has been observed in the RAS-MAPK pathway and low bone mineral density has already been described in this population.

Joint lesions and their evolution remain poorly described in the literature. The early pediatric diagnosis of Noonan's syndrome is important in detecting multiple organ damage. Early management should improve joint functional prognosis.

The objective of this work is therefore to evaluate the frequency and type of these events in the French pediatric population and to compare patients with and without these disorders, and to observe the proposed treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≤ 20 years at the time of diagnosis
* Noonan syndrome confirmed by van der Burgt score
* At least one consultation in the participating center

Exclusion Criteria:

* Patient > 20 years old at the time of diagnosis
* Absence of diagnostic criteria for van der Burgt's Noonan syndrome
* Other rasopathies
* Genetic mutations of MEK1, MEK2 and HRAS (which are associated with cardi-faci-cutaneous syndrome and Costello syndrome)
* Refusal of participation in the study

Ages: 0 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: French pediatric population, followed for a syndrome of Noonan clinically confirmed by the criteria of Van der Burgt.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2020-03-28 (Actual); Study Completion 2020-03-28 (Actual)

PRIMARY OUTCOMES:
Description of joint and hematologic disorders in patients with Noonan syndrome clinically confirmed by Van der Burgt criteria. | Inclusion (Day 0)
  Joint disorders
Description of joint and hematologic disorders in patients with Noonan syndrome clinically confirmed by Van der Burgt criteria. | Inclusion (Day 0)
  hematologic disorders

SECONDARY OUTCOMES:
Comparison of patients with and without joint involvement. | Inclusion (Day 0), Each year
  Comparison of patients with and without joint involvement.
Comparison of patients with and without joint involvement. | Inclusion (Day 0), Each year
  Evolution of joint damage with and without treatment.

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CHRU de Brest, Brest
  - CHU de Caen, Caen
  - CHU de Nantes, Nantes
  - CHU de Toulouse, Toulouse